CLINICAL TRIAL: NCT03856294
Title: A Placebo-controlled Study on the Effect of Rikkunshito on Gastric Accommodation and Nutrient Volume Tolerance, Quantified by Intragastric Pressure Monitoring During Intragastric Nutrient Infusion, in Functional Dyspepsia
Brief Title: The Effect of Rikkunshito on Gastric Accommodation and Nutrient Volume Tolerance in Functional Dyspepsia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Tsumura and Company, Tokyo, Japan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Rikkunshito1
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Dyspepsia
Keywords: gastric motility; functional dyspepsia; functional dyspepsia symptoms
MeSH Terms: conditions — Dyspepsia | interventions — liu-jun-zi-tang

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rikkunshito (Experimental): Rikkunshito: 2,5g dissolved in 200 mL lukewarm water, three times daily, 30min before meal intake
  Interventions: Drug: Rikkunshito
- Placebo (Placebo Comparator): Placebo: 2,5g dissolved in 200 mL lukewarm water, three times daily, 30min before meal intake
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Rikkunshito — Rikkunshito, 2,5g dissolved in 200 mL lukewarm water, three times daily, 30min before meal intake
  Other Names: TJ-43
  Arms: Rikkunshito
Drug: Placebos — Placebo, 2,5g dissolved in 200 mL lukewarm water, three times daily, 30min before meal intake
  Arms: Placebo

SUMMARY:
Functional dyspepsia (FD) is a common chronic gastrointestinal (GI) disorder. Rikkunshito, a traditional Japanese Kampo medicine, has shown efficacy in improving FD symptoms in controlled trials in Japan. Its putative benefit for European patients has never been investigated. Further, its exact mechanism of action is incompletely elucidated. This study aimed to examine the effect of rikkunshito on gastric motility and GI symptom perception in FD in a randomized, placebo-controlled, cross-over study. Intragastric pressure (IGP) was assessed using high-resolution manometry as an indirect measurement of gastric accommodation and gastric motility.

DETAILED DESCRIPTION:
This randomized, placebo-controlled, double-blind, cross-over study had a total duration of 14 weeks, consisting of a two-week run-in period, two treatment phases of four weeks each and a four-week washout period separating the treatment phases to prevent carry-over effects. Study visits were held at baseline (screening) and after the run-in period, treatment phases and washout period.

To assess the effect of rikkunshito on intragastric pressure as an indirect measure for gastric motility, high-resolution manometry (HRM) was performed after the run-in period and after both treatment phases. During intragastric pressure measurement, a nutrient tolerance test was performed and symptom questionnaires were completed. Throughout the entire study, patients scored their gastrointestinal symptoms on a daily basis in the Leuven Postprandial Distress Scale (LPDS) diary. In addition, questionnaires on gastrointestinal symptoms and psychosocial state were completed each study visit.

Safety measures performed each study visit included blood pressure, heart rate and weight assessment, performing an electrocardiogram, adverse event evaluation and physical examination. Furthermore, blood samples were collected during screening and after each treatment phase to check liver and kidney function. Serum levels of potassium, creatine kinase, aspartate aminotransferase, alanine transaminase, alkaline phosphatase and gamma- glutamyltransferase were assessed. Women of childbearing potential were asked to do a pregnancy test before study enrollment and before each treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with FD-postprandial distress syndrome subtype diagnosis as per Rome IV
2. Patients must provide witnessed written informed consent prior to any study procedures being performed
3. Patients aged between 18 and 75 years inclusive
4. Male or female patients. Women of child-bearing potential agree to apply during the entire duration of the trial a highly effective method of birth control, which is defined as those which result in a low failure rate (i.e., less than 1% per year) when used constantly and correctly such as implants, injectables, combined oral contraceptive method, or some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. Women of non-childbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or postmenopausal with at least 2 year without spontaneous menses.
5. Patients who are capable to understand the study and the questionnaires, and to comply with the study requirements

Exclusion Criteria:

1. Patients with any condition which, in the opinion of the investigator, makes the patient unsuitable for entry into the study
2. Patients with an active major psychiatric condition (depression, anxiety disorder, alcohol or substance abuse). However, patients who are taking a stable dose of a single antidepressant (with the exception of amitryptiline and mirtazapine which are forbidden) during the last 3 months are eligible.
3. Females who are pregnant or lactating. Females who refuse to take appropriate contraception at the time of informed consent.
4. Men who want to donate sperm during the study and during the 4 weeks after stopping Rikkunshito.
5. Patients who received treatment for Helicobacter Pylori (HP) eradication during the last 3 months. Patients who are HP positive may enter the study provided that their endoscopy is negative. If HP status is unknown, determination of HP status will be done during run-in.
6. Patients suffering from diabetes type 1 or type 2.
7. Patients taking drugs affecting the gut secretion, mucosal integrity (non-steroidal anti-inflammatory drugs (NSAIDs), with an exception for aspirin at cardioprotective dose of max 125 mg daily), motility, and/or sensitivity. Patients taking proton pump inhibitors (PPIs) are eligible provided that FD is predominant and heartburn limited to maximum two episodes of mild intensity per week.
8. Patients with coronary heart disease, arrhythmias or taking concomitant drugs capable to prolong the QT.
9. Patients taking concomitant drugs able to induce drug-drug interaction (P450), Concomitant drugs interacting substantially with the different fractions of cytochromes (CYP3A4 and others) and with strong protein binding (Albumine, i-globulins, acid glycoproteins) are excluded.
10. Patients with a significant renal [serum creatinine >2 x upper limit of normal (ULN)], hepatic [alanine transaminase (ALT), aspartate transaminase (AST), gamma glutamyltransferase (GGT), bilirubin >2 x ULN], cardiovascular, pulmonary, endocrine, metabolic or haematological condition.
11. Patients with known hypersensitivity to the Ginseng or Ginger.
12. Patients with confirmed gastro-intestinal disease.
13. Patients with former digestive surgery affecting upper gut motility.
14. Patients affected by concomitant extra-digestive disease responsible for digestive symptoms.
15. Patients presenting with predominant symptoms of irritable bowel syndrome (IBS).
16. Patients presenting symptoms of epigastric pain syndrome (EPS) several times a week, not related to meals, according to Rome III questionnaire (score 5 or higher on question 10, in combination with clinical judgement).
17. Patients presenting daily symptoms of nausea syndrome, not related to meals, on Rome III questionnaire (score 6 on question 6 or score 5 or higher on question 9).
18. Patients presenting vomiting more than one day a month.
19. Patients presenting daily symptoms of Excessive belching according to Rome III questionnaire (score 6 on question 19, in combination with clinical judgement).
20. Patients presenting predominant gastro-esophageal reflux disease (GERD) (3 "yes" by GERD questionnaire, in combination with clinical judgement).
21. Patients not willing to take ultraviolet protective measures or patients at increased risk for phototoxicity (use of drugs like tetracyclins, amiodarone, sulphonamides, quinolones).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Gastric pressure | Gastric pressure was measured until 2 hours after the start of the liquid meal. Liquid meal started 30 minutes after rikkunshito/placebo intake
  Contractions of the stomach and relaxation of the stomach upon food intake

SECONDARY OUTCOMES:
Gastrointestinal symptoms during gastric pressure measurement | every 5 minutes, up to 2 hours after administration of the liquid meal
  Change in subjective gastrointestinal symptom scores measured by visual analogue scale of 100 mm
Gastrointestinal symptoms during treatment period | On a daily basis throughout the 4-week treatment arms
  change in subjective gastrointestinal symptom scores throughout both treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No